CLINICAL TRIAL: NCT00151970
Title: A Phase IIB, Randomized, Double-blind, Multi-Center, Placebo-Controlled, Dose-Optimization, 3-way Cross-Over, Analog Classroom Study to Assess the Efficacy, Duration of Effect, Tolerability and Safety of 4- and 6- Hour Wear Times of Methylphenidate Transdermal System (MTS) in Pediatric Subjects Aged 6-12 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Efficacy, Safety and Tolerability of SPD485 in Children Aged 6-12 Diagnosed With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Collaborators: Noven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD485-304
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Methylphenidate Transdermal System (Active Comparator): The duration of MTS patch wear was 9 hours per day. A new patch was applied each morning upon awakening.
  Interventions: Drug: Methylphenidate Transdermal System
- Placebo (Placebo Comparator): The duration of placebo patch wear was 9 hours per day. A new patch was applied each morning upon awakening.
  Interventions: Drug: Placebo
- Concerta (Active Comparator): CONCERTA® is available in doses of 18mg, 27mg, 36mg, 54mg, and 72mg tablets daily
  Interventions: Drug: Concerta

INTERVENTIONS:
Drug: Methylphenidate Transdermal System — MTS 10mg/12.5cm2, 15mg/18.75cm2, 20mg/25cm2, and 30mg/37.5cm2 patch sizes
  Other Names: MTS
  Arms: Methylphenidate Transdermal System
Drug: Placebo — Placebo patch 10mg/12.5cm2, 15mg/18.75cm2, 20mg/25cm2, and 30mg/37.5cm2 patch sizes applied daily
  Other Names: Sham Treatment
  Arms: Placebo
Drug: Concerta — CONCERTA® is available in doses of 18mg, 27mg, 36mg, 54mg, and 72mg tablets daily
  Other Names: Methylphenidate HCL
  Arms: Concerta

SUMMARY:
This study will assess the efficacy, duration of effect, tolerability and safety of 4- and 6- hour wear times of SPD485 in 6-12 year old subjects diagnosed with ADHD.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a psychiatric disorder characterized by 3 main symptoms: inattention, hyperactivity and impulsivity. This study will assess the efficacy, duration of effect, tolerability and safety of 4- and 6- hour wear times of SPD485 in 6-12 year old subjects diagnosed with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have primary diagnosis of ADHD
* Females of childbearing potential must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test
* Subject has an IQ score of >_ 80
* Subject is able to complete as least the Basic Test of the PERMP assessment

Exclusion Criteria:

* Subject has a comorbid psychiatric diagnosis such as Axis II disorders or severe Axis I disorders
* Subject is taking Strattera(r)
* Subject has a recent history of suspected substance abuse or dependence disorder

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2005-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
SKAMP deportment rating scale | Week 8

SECONDARY OUTCOMES:
PERMP age-adjusted math test | Week 8
Clinician-rated ADHD-RS-IV | Week 8
CGI-I | Week 8
Parent Global Assessment | Week 8
Connors' Parent Rating Scale | Week 8
ADHD Impact Module-Children | Week 8
SKAMP-total and inattention subscales | Week 8

REFERENCES:
- [Background] Wilens TE, Boellner SW, Lopez FA, Turnbow JM, Wigal SB, Childress AC, Abikoff HB, Manos MJ. Varying the wear time of the methylphenidate transdermal system in children with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2008 Jun;47(6):700-708. doi: 10.1097/CHI.0b013e31816bffdf. PMID 18434918
- [Derived] Frazier TW, Weiss M, Hodgkins P, Manos MJ, Landgraf JM, Gibbins C. Time course and predictors of health-related quality of life improvement and medication satisfaction in children diagnosed with attention-deficit/hyperactivity disorder treated with the methylphenidate transdermal system. J Child Adolesc Psychopharmacol. 2010 Oct;20(5):355-64. doi: 10.1089/cap.2009.0092. PMID 20973706
- [Derived] Manos M, Frazier TW, Landgraf JM, Weiss M, Hodgkins P. HRQL and medication satisfaction in children with ADHD treated with the methylphenidate transdermal system. Curr Med Res Opin. 2009 Dec;25(12):3001-10. doi: 10.1185/03007990903388797. PMID 19849639
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html